CLINICAL TRIAL: NCT05458674
Title: A Phase II Study of the Safety, Tolerability and Antitumor Activity of Tucatinib in Combination With Eribulin and Trastuzumab in Patients With Pretreated Unresectable Locally Advanced or Metastatic HER2+ Breast Cancer
Brief Title: Tucatinib+Trastuzumab+Eribulin in HER2+ MBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Criterium, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02AB21-TucErBit
Record Dates: First submitted 2022-06-27; First posted 2022-07-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Pretreated Unresectable Locally Advanced or Metastatic HER2+ Breast Cancer
Keywords: Pretreated Unresectable locally advanced or metastatic HER2+ breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib; eribulin; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tucatinib/Eribulin/Trastuzumab (Experimental): * The initial dose of trastuzumab will be given as a loading dose of 8 mg/kg intravenously (IV), unless trastuzumab was administered within the prior 4 weeks, then the initial dose of trastuzumab will be administered at a dose of 6 mg/kg. Each trastuzumab dose is given once every 21 days, except in specific circumstances where it may be given weekly to compensate for modifications in treatment schedule
  * Tucatinib 300 mg orally twice daily (PO BID) every day (Days 1-21) of each 21-day cycle using a modified schedule of events. Subcutaneous trastuzumab is given only once every three weeks as there is no allowance for weekly dosing.
  * Eribulin will be given at a dose of 1.1 mg/M2 intravenously over a 2-5 minute period on days 1 and 8 of each 21-day cycle.
  Interventions: Drug: Tucatinib; Drug: Eribulin; Drug: Trastuzumab

INTERVENTIONS:
Drug: Tucatinib — taken orally
  Other Names: TUKYSA
Drug: Eribulin — taknen intravenously
  Other Names: HALAVEN
Drug: Trastuzumab — taken intravenously
  Other Names: HERCEPTIN

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the three-drug combination of tucatinib, trastuzumab, and eribulin in patients with de novo and recurrent unresectable metastatic HER-2/neu positive breast cancer as assessed by ORR, PFS and OS after prior treatment with a taxane, trastuzumab, and T-DM1.

DETAILED DESCRIPTION:
In view of the potency of tucatinib for the treatment of brain metastases and its modest toxicity, it is important to evaluate the combination of this drug with other established anti-HER2 therapies. There remains a need to evaluate the efficacy of tucatinib with additional active agents in this area. Given the demonstrated activity of eribulin in metastatic breast cancer in general and in her2 positive disease combined with trastuzumab in particular, this study proposes to evaluate the safety and efficacy of the three-drug combination of eribulin, trastuzumab, and tucatinib. It is also important to ascertain the activity of this combination in patients who have previously received tucatinib, as little is known about whether resistance to tucatinib plus one chemotherapy drug confers resistance to tucatinib with a different partner drug.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed HER2+ breast carcinoma, with HER2+ defined by in situ hybridization (ISH) or fluorescence in situ hybridization (FISH) or immunohistochemistry (IHC)
2. Have received previous treatment with trastuzumab deruxtecan in the metastatic setting or have recurred within 6 months of receiving this treatment in the adjuvant or neoadjuvant setting. Prior taxane, capecitabine and T-DM1 are not required. Prior tucatinib therapy is allowed. Patients for whom Trastuzumab is contraindicated are not permitted. Have progression of unresectable locally advanced or metastatic breast cancer after last systemic therapy (as confirmed by site investigator),or be intolerant of last systemic therapy.
3. Have measurable or non-measurable disease assessable by RECIST 1.1
4. Be at least 18 years of age at time of consent.
5. Have Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0,1 or 2
6. Have a life expectancy of at least 6 months, in the opinion of the site investigator.
7. Have adequate hepatic function as defined by the following:

   1. Total bilirubin ≤1.5 X upper limit of normal (ULN), except for patients with known Gilbert's disease, who may enroll if the conjugated bilirubin is ≤1.5 X ULN
   2. Transaminases [aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT)] ≤ 2.5 X ULN (≤ 5 X ULN if liver metastases are present)
8. Have adequate baseline hematologic parameters as defined by:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 103/µL
   2. Platelet count ≥ 100 x 103/µL; patients with stable platelet count from 75- 100 x 103/µL may be included with approval from medical monitor,
   3. Hemoglobin ≥ 9 g/dL
   4. In patients transfused before study entry, transfusion must be ≥ 14 days prior to start of therapy to establish adequate hematologic parameters independent from transfusion support,
9. Have creatinine clearance ≥ 50 mL/min as calculated per institutional guidelines or, in patients ≤ 45 kg in weight, a serum creatinine within institutional normal limits,
10. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 X ULN unless on medication known to alter INR and aPTT. (Note: Warfarin and other coumarin derivatives are prohibited.)
11. Have left ventricular ejection fraction (LVEF) ≥ 50% as assessed by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA) documented within 4 weeks prior to first dose of study treatment.
12. If female of childbearing potential, must have a negative result of serum or urine pregnancy test performed within 7 days prior to first dose of study treatment. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post- menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

    NOTE: Postmenopausal patients with known β-HCG secreting tumors may be eligible when β-HCG-based urine or serum pregnancy tests yield false positive if they meet the definition of postmenopausal state and have a negative uterine ultrasound
13. Women of childbearing potential (as defined above) and men with partners of childbearing potential must agree to use a highly effective birth control method, i.e., methods that achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal); progestogen- only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable); intrauterine device; intrauterine hormone-releasing system; bilateral tubal occlusion/ligation; vasectomized partner; or sexual abstinence. Male patients with partners of childbearing potential must use barrier contraception. All study patients should practice effective contraception, as described above, starting from the signing of informed consent until 7 months after the last dose of study medication or investigational medicinal product.
14. Patient must provide signed informed consent per a consent document that has been approved by an institutional review board or independent ethics committee (IRB/IEC) prior to initiation of any study-related tests or procedures that are not part of standard-of-care for the patient's disease.
15. Patients must be willing and able to comply with study procedures.

CNS Inclusion - Based on screening contrast brain magnetic resonance imaging (MRI), patients must have one of the following:

1. No evidence of brain metastases
2. Untreated brain metastases not needing immediate local therapy. For patients with untreated CNS lesions > 2.0 cm on screening contrast brain MRI, discussion with and approval from the medical monitor is required prior to enrollment,
3. Previously treated brain metastases a. Brain metastases previously treated with local therapy may either be stable since treatment or may have progressed since prior local CNS therapy, provided that there is no clinical indication for immediate re-treatment with local therapy in the opinion of the site investigator, b. Patients treated with CNS local therapy for newly identified lesions found on contrast brain MRI performed during screening for this study may be eligible to enroll if all of the following criteria are met: i. Time since whole brain radiation therapy (WBRT) is ≥ 21 days prior to first dose of study treatment, time since stereotactic radiosurgery (SRS) is ≥ 7 days prior to first dose of study treatment, or time since surgical resection is ≥ 28 days, ii. Other sites of disease assessable by RECIST 1.1 are present, iii. Relevant records of any CNS treatment must be available to allow for classification of target and non-target lesions

Exclusion Criteria:

1. Have previously been treated with eribulin for metastatic disease (except in cases where eribulin was given for ≤ 21 days and was discontinued for reasons other than disease progression or severe toxicity)
2. History of exposure to the following cumulative doses of anthracyclines:

   1. Doxorubicin > 360 mg/m2
   2. Epirubicin > 720 mg/m2
   3. Mitoxantrone > 120 mg/m2
   4. Idarubicin > 90 mg/m2
   5. Liposomal doxorubicin (e.g. Doxil, Caelyx, Myocet) > 550 mg/m2
3. History of allergic reactions to trastuzumab, eribulin, or compounds chemically or biologically similar to tucatinib, except for Grade 1 or 2 infusion related reactions to trastuzumab that were successfully managed, or known allergy to one of the excipients in the study drugs
4. Have received treatment with any systemic anti-cancer therapy (including hormonal therapy), non-CNS radiation, or experimental agent ≤ 3 weeks of first dose of study treatment or are currently participating in another interventional clinical trial. An exception for the washout of hormonal therapies is gonadotropin releasing hormone (GnRH) agonists used for ovarian suppression in premenopausal women, which are permitted concomitant medications.
5. Have any toxicity related to prior cancer therapies that has not resolved to ≤ Grade 1, with the following exceptions:

   1. alopecia and neuropathy, which must have resolved to ≤ Grade 2; and
   2. congestive heart failure (CHF), which must have been ≤ Grade 1 in severity at the time of occurrence, and must have resolved completely.
   3. anemia, which must have resolved to ≤ Grade 2
6. Have clinically significant cardiopulmonary disease such as:

   1. ventricular arrhythmia requiring therapy,
   2. uncontrolled hypertension (defined as persistent systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 100 mm Hg on antihypertensive medications)
   3. any history of symptomatic CHF
   4. severe dyspnea at rest (CTCAE Grade 3 or above) due to complications of advanced malignancy
   5. hypoxia requiring supplementary oxygen therapy except when oxygen therapy is needed only for obstructive sleep apnea.
   6. Presence of Grade 2 or greater QTc prolongation on screening ECG.
   7. conditions potentially resulting in drug-induced prolongation of the QT interval or torsade de pointes:

   i. Congenital or acquired long QT syndrome. ii. Family history of sudden death iii. History of previous drug induced QT prolongation iv. Current use of medications with known and accepted associated risk of QT prolongation
7. Have known myocardial infarction or unstable angina within 6 months prior to first dose of study treatment.
8. Have chronic active Hepatitis B or Hepatitis C or have other known chronic liver disease.
9. Are known to be positive for human immunodeficiency virus (HIV)
10. Are pregnant, breastfeeding, or planning a pregnancy.
11. Require therapy with warfarin or other coumarin derivatives (non-coumarin anticoagulants are allowed)
12. Have inability to swallow pills or significant gastrointestinal disease which would preclude the adequate oral absorption of medications.
13. Use of a strong CYP3A4 or CYP2C8 inhibitor within 5 half-lives of the inhibitor, or use of a strong CYP3A4 or CYP2C8 inducer within 5 days prior to first dose of study treatment
14. Unable for any reason to undergo contrast MRI of the brain.
15. Have any other medical, social, or psychosocial factors that, in the opinion of the investigator, could impact safety or compliance with study procedures.
16. Have evidence within 2 years of the start of study treatment of another malignancy that required systemic treatment.

CNS Exclusion - Based on screening brain MRI, patients must not have any of the following:

1. Any untreated brain lesions > 2.0 cm in size, unless discussed with medical monitor and approval for enrollment is given.
2. Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of > 2 mg of dexamethasone (or equivalent). However, patients on a chronic stable may be eligible with discussion and approval by the medical monitor.
3. Any brain lesion thought to require immediate local therapy, including (but not limited to) a lesion in an anatomic site where increase in size or possible treatment-related edema may pose risk to patient (e.g., brain stem lesions). Patients who undergo local treatment for such lesions identified by screening contrast brain MRI may still be eligible for the study based on criteria described under CNS inclusion criteria 19b.
4. Have poorly controlled (> 1/week) generalized or complex partial seizures, or manifest neurologic progression due to brain metastases notwithstanding CNS-directed therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of tucatinib in combination with eribulin and trastuzumab in patients with unresectable or recurrent metastatic HER2+ breast cancer who have had prior treatment with trastuzumab, and trastuzumab deruxtecan. | 2 years
  Incidence of adverse events and serious adverse events. Rate of grade 3 -4 toxicity, incidence of dose limiting toxicities, incidence of dose holding, dose reductions, and discontinuations of any and/or all of the three treatment agents. Incidence of cardiac and pulmonary complications.
Evaluate the relative toxicity/tolerability of these therapeutic agents when used in combination in this patient cohort | 2 years
  Rate of grade 3 -4 toxicity, incidence of dose limiting toxicities, incidence of dose holding, dose reductions, and discontinuations of any and/or all of the three treatment agents

SECONDARY OUTCOMES:
Evaluate efficacy against HER2 + metastatic breast cancer | 2 years
  Overall response rate (ORR) and progression-free survival (PFS) will be assessed per RECIST 1.1 criteria
Evaluate efficacy against CNS disease | 2 years
  progressive disease will be assessed per RANDO-BM criteria
Efficacy in patients who have had prior tucatinib | 2 years
  Assessed per Overall survival and Progression Free survival in patients who have received prior tucatinib therapy
Efficacy in treating CNS disease | 2 years
  Assessed per Overall survival and Progression Free survival in patients with CNS disease

CONTACTS AND LOCATIONS:
Overall Officials: Hank Kaplan, MD, Principal Investigator — henry.kaplan@swedish.org
Locations (6):
- United States (6):
  - University of Colorado, Aurora, Colorado
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Swedish Cancer Institute, Issaquah, Washington
  - Cancer Care Northwest, Spokane Valley, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided